CLINICAL TRIAL: NCT06272708
Title: Preliminary Exploration of Thromboelastography in the Monitoring of Anticoagulation in Maintenance Hemodialysis Patients
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Renhua Lu, Chief Physician, RenJi Hospital
Other Study IDs: IIT-2023-0356
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Thromboelastography; Hemodialysis; Anticoagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objectives: To investigate the role of thromboelastography parameters (R, K, Angle, MA) in monitoring anticoagulation in maintenance hemodialysis (MHD) patients.

Subjects: Two hundred stable MHD patients. Methods: An observational study. Primary outcome: Relationship between thromboelastography parameter R Value and coagulation of hemodialysis circuit and dialyzer.

Secondary outcome: Relationship between thromboelastography parameters (K Value, Angle and MA) and coagulation of hemodialysis circuit and dialyzer.

ELIGIBILITY:
Inclusion Criteria:

1. male or female patients aged over 18 years
2. stable patients undergoing maintenance hemodialysis treatment for at least 3 months
3. signed informed consent form

Exclusion Criteria:

1. concomitant with severe diseases such as active malignancy, severe liver diseases, systemic infection, etc.
2. planned or ongoing pregnancy or lactation
3. unsuitable for inclusion in this study after assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stable patients undergoing maintanence hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
thromboelastography parameter R value | 2 hours after hemodialysis began
  Relationship between thromboelastography parameter R value and coagulation of hemodialysis circuit and dialyzer

SECONDARY OUTCOMES:
thromboelastography parameter K value | 2 hours after hemodialysis began
  Relationship between thromboelastography parameter K value and coagulation of hemodialysis circuit and dialyzer
thromboelastography parameter Angle | 2 hours after hemodialysis began
  Relationship between thromboelastography parameter Angle and coagulation of hemodialysis circuit and dialyzer
thromboelastography parameter MA | 2 hours after hemodialysis began
  Relationship between thromboelastography parameter MA value and coagulation of hemodialysis circuit and dialyzer

CONTACTS AND LOCATIONS:
Overall Officials: Yiwei Shen, MD, Principal Investigator — RenJi Hospital; Renhua Lu, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China